CLINICAL TRIAL: NCT05135507
Title: The Effective Parenting Program (EPP): An Integrated Stress Reduction and Parenting Intervention for Families of Children With Developmental Disabilities
Brief Title: The Effective Parenting Program (EPP)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 - unable to recruit any participants
Sponsor: Double S Instructonal Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPPPhaseI
Record Dates: First submitted 2021-10-28; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Parent-Child Relations

STUDY DESIGN:
Intervention Model Description: Within subject pre and posttest design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- An interactive stress reduction and behavioral parent training program (Experimental): This feasibility evaluation will track and analyze individual program usage and examine changes in parents' psychological flexibility, parents' stress, parenting self-efficacy, parents' mindfulness and child behavior in a within subject pretest and posttest design with 50 parents of children who have DD
  Interventions: Behavioral: An integrated parenting intervention for families of children with developmental disabilities

INTERVENTIONS:
Behavioral: An integrated parenting intervention for families of children with developmental disabilities — Deliver three training modules to parent and track program usage, psychological flexibility, parents' stress, parents mindfulness, and child behavior

SUMMARY:
The Phase I objective is to determine the feasibility of the EPP program by examining user responses to the first three units of EPP's nine interactive training modules. This feasibility evaluation will track and analyze individual program usage and examine changes in parents' psychological flexibility, parents' stress, parenting self-efficacy, parents' mindfulness and child behavior in a within subject pretest and posttest design with 50 parents of children who have DD. Qualifying parents will complete a baseline assessment and then be directed to our online learning platform to complete the interactive learning activities. This test of the Phase I prototype is intended to approximate the conditions under which the complete product will be marketed and used.

DETAILED DESCRIPTION:
Parents who have children with developmental disabilities (DD) commonly experience high levels of stress related to child behavior problems and contextual issues related to the child's disability that can have a detrimental effect on their parenting. Current stress management programs for this population of parents often do not lead to a reduction in children's behavior problems and Behavioral Parent Training programs (BPT) do not always lead to a reduction in stress. Interventions that combine the two approaches are more effective, providing substantial benefits to both parent and child. The central goal of this project is to create an online, interactive stress reduction and BPT program: The Effective Parenting Program (EPP): An Integrated Parenting Intervention for Families of Children with Developmental Disabilities. The investigators propose three Specific Aims with the primary aims of reducing parents' stress and strengthening parents' parenting efficacy and psychological flexibility. The investigators secondary aims are designed to answer questions regarding (a) the influence of changes in parents' efficacy and psychological flexibility on child behavior and (b) the role of parents' attention to and awareness of present moment experiences. This work is significant because it will provide resources for an underserved population - parents of children with DD -- who experience frequent stress with the challenges of raising a child with DD and who may lack basic behavioral parenting skills. Moreover, the proposed program has the potential to broadly impact the way supports are delivered to parents of children with DD by adding an integrated, efficacious intervention that overcomes common barriers to parental participation (time, finances, and availability). From a public health perspective, this approach is ideally structured to meet the needs of this population of parents who are in need of easy to implement and cost effective support and training.

Upon completion in Phase II, parents will have access to a complete EPP program, designed to help parents cope with stress more effectively and strengthen their behavioral parenting skills. The program will provide parents with engaging, interactive content, including: tools for monitoring progress, text prompts and incentives to motivate behavior change, a mechanism for the sharing of social support, guidance in setting effective value-based goals, strategies for reducing stress, and training in evidence-based parenting skills. The EPP program will be available on a mobile website that can be accessed by smart phones, tablets and computers and will provide realistic situational videos vignettes, workbook exercises and a discussion forum to help parents deal effectively with stress and challenging behaviors. In Phase I of this project, the investigators will determine the feasibility of the program by examining primary and secondary outcomes related to a prototype of the EEP program.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children with developmental disabilities having a child with Developmental Disabilities who lives at home (50% of parents will have a child with autism and 50% will have a child with intellectual disabilities,
* Must have access to a phone that can receive text messages and an Internet connection,
* Stress levels being elevated (i.e., greater than .5 standard deviations above the normative data mean score) on a 12 item Parental distress sub scale of the Parenting Stress Index- short form.

Exclusion Criteria:

* Parents of children without a developmental disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Acceptance and Action Questionnaire II (AAQ-II) | Change from baseline acceptance at five weeks post
  Measures the extent to which individuals were able to experience upsetting or difficult thoughts, feelings and emotions without trying to suppress or avoid them and to take valued action, even in the midst of difficult internal experiences.It is comprised of 7 items rating scale with 1=never true and 7= always true
Parental Stress Scale | Change from baseline parental stress at five weeks post
  The PSS consists of 18 items that measure the levels of stress parents experience as a result of having children. Parents respond by indicating the extent that they agree or disagree with each statement on a 5 point scale.5 point scale; strongly disagree, disagree, undecided, agree, strongly agree
Child Adjustment and Parent Efficacy Scale(CAPES) | Change from baseline child adjustment and parental self-efficacy at five weeks post
  the CAPES consists of a 30-item intensity scale with two subscales measuring child behavior problems, child prosocial behavior and emotional maladjustment and a 20-item self-efficacy scale assessing parents parent's self-efficacy in handling specific child problem behaviors.4 point rating scale with 0=not at all and 3=very much

SECONDARY OUTCOMES:
Mindful Attention Awareness Scale (MAAS) | Change in attention and awareness from Baseline at five weeks post
  This 18 item instrument measures participant's tendency to be attentive to and aware of present moment experiences in daily life.6 point scale
  1= almost always and 6 = almost never
Parent Social Validity Questionnaire (PSVQ) | five weeks post
  This 6-item survey will assess parent perceptions of the materials and the extent to which they have been practicing the techniques they had learned. Parents will indicate the extent to which they agree with each item on a 7-point Likert scale. The items are rated on a five point scale -- 1=strongly agree to 5= strongly disagree.6 items consisting of a 5 item rating scales items 1-5 with 1=none and 6 = very much And item 6 asks them to check of a list of 5 barriers to doing the program